CLINICAL TRIAL: NCT06540495
Title: Virtual Personalized Exercise Program for Subjects With Lung Cancer: a Feasibility Study
Brief Title: Virtual Personalized Exercise Program for Lung Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Salaso (Unknown); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-0199
Record Dates: First submitted 2024-07-18; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Exercise
MeSH Terms: conditions — Lung Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: Prospective, Single Arm (Three Cohorts), Open Label, Feasibility study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm Study (Experimental): Cohort A: Peri-operative (subjects starting neoadjuvant chemotherapy or within 4-8 weeks after curative-intent thoracic surgery which could be segmentectomy, lobectomy of pneumonectomy), irrespective of adjuvant treatment - expected recruitment: 15 subjects
  Cohort B: Subjects Subjects starting definitive chemotherapy and radiation for locally advanced lung cancer- expected recruitment: 15 subjects
  Cohort C: Subjects with stage IV metastatic non-small cell lung cancer irrespective of type of treatment - expected recruitment: 30 subjects
  Interventions: Behavioral: Salaso Virtual Exercise Program

INTERVENTIONS:
Behavioral: Salaso Virtual Exercise Program — Salaso is a digital health technology company that has online, mobile and telehealth solutions enabling providers to 'prescribe' evidence-based exercise programs for patients to complete virtually.

SUMMARY:
This is a prospective study providing lung cancer subjects at R.J. Zuckerberg Cancer Center with a customized exercise program provided by Salaso, with the goal of improving functional status and outcomes. This study will assess the feasibility and usability of a virtual exercise platform designed for lung cancer subjects. Subjects will be referred to physical therapy and rehabilitation medicine doctors for evaluation and enrolment in a virtual exercise program tailored specifically to their needs. The virtual exercise program will be available on a digital platform accessible through a personal device. Subjects will undergo a pulmonary function test if not previously completed within 3 months of signing consent, a Six minute walk test (6MWT) and the Sit to Stand Test (STS) at the start and end of the 12- month program. Subjects will also be asked to complete quality of life FACT-L and the Patient Satisfaction questionnaires at 1 month, 3-months, 6-months, and 12-months. Patient satisfactions questionnaires include the System Usability Scale, Net Promotor Score (NPS), and the Technology Acceptance Model. Physicians will also complete a provider satisfaction questionnaire at 1 month, 6 months, 12 months, and 24 months from the time their first patient is enrolled. Subject participation in the trial will last 12 months from the time the subject starts utilizing the platform. If we find that the platform is accepted by subjects and is found to be feasible, a future randomized study will be developed to follow.

Eligibility criteria (note that subjects will be allowed to be enrolled in the program as long as it is within 3 weeks of starting treatment):

i. Subjects with Non-small cell lung cancer who belong to any of the three cohorts below ii. Have an ECOG PS of 0-2 iii. Can provide informed consent iv. Can engage in a virtual exercise platform v. Commit to all study procedures as per protocol vi. Are deemed appropriate for virtual exercise program by the PM&R team

The following three cohorts of subjects will be eligible for this feasibility study:

1. Cohort A: Peri-operative (subjects starting neoadjuvant chemotherapy or within 4-8 weeks after curative-intent thoracic surgery which could be segmentectomy, lobectomy of pneumonectomy), irrespective of adjuvant treatment).

1. Expected recruitment - 15 subjects
2. Cohort B: Subjects starting definitive chemotherapy and radiation for locally advanced lung cancer.

1. Expected recruitment - 15 subjects

3. 3. Cohort C; Subjects with stage IV metastatic non-small cell lung cancer irrespective of type of treatment.

1. Expected recruitment - 30 subjects

DETAILED DESCRIPTION:
Cancer as a chronic disease: Cancer is now considered a chronic disease and the number of cancer survivors is estimated to be more than 22 million individuals in the United States by 2030.[1]

Cancer and exercise: As opposed to chronic conditions such as heart disease, diabetes, and pulmonary disease where exercise has been recommended for decades, exercise recommendations for oncologists has been slow to evolve. However, exercise and rehabilitation interventions are known to benefit cancer survivors. Interestingly, research has been shown that the risk of developing cancer can be reduced by exercising a minimum of 3 - 5 hours per week, reducing the risk of breast cancer by 15 to 20%, decreasing the risk of colorectal cancer by 19-24%, gastric cancer by 19%, kidney cancer by 23%, and esophageal cancer by 21%.[2, 3] While we know a lot about exercise beneficial effects on the heart and skeletal muscle, studies are emerging on its effects on other organs where cancer cells grow including breast, prostate, colon, pancreas, kidney, liver and lung. Exercise can also play a role in cancer treatment by reducing treatment-related toxic and side effects and enhancing the curative effects of other treatments.[2] For those undergoing active cancer treatment, exercise has proven benefits. For example, breast cancer subjects treated with aromatase inhibitors develop decreased cognitive ability and lower bone mass.[2] Exercise is thought to prevent cognitive impairments caused by estrogen deficiency. Similarly, for prostate cancer, physical exercise can improve androgen-deprivation therapy. The most reported issues for cancer survivors are physical problems (muscle mass reduction, pain, and fatigue) and psychosocial problems (depression, cognitive decline, and fear of recurrence) and increased risk of developing secondary comorbidities such as cardiovascular disease.[4] Physical exercise has been shown to improve fatigue related to cancer treatment, likely by mitigating oxidative stress and reducing hormone stimulation. Additionally, those who exercise post-colon resection have a 50% reduction in disease-free survival when comparing 18 to 27 metabolic equivalent task (MET)-hours per week versus less than three MET-hours per week.[5] Observational cohort studies show that subjects who have high physical activity after diagnosis have lower risk of disease recurrence and cancer mortality.[6] Randomized clinical trials have also validated that physical activity interventions both mitigate cancer-impaired quality of life and improve outcomes for cancer survivors. One in ten cancer deaths have been attributed to lack of physical activity.[7] And, a recent meta-analysis of 38,560 cancer survivors demonstrated a 37% lower relative risk of dying from cancer for the most active compared with the least active subjects (HR: 0.63; 95% CI: 0.54-0.73).[8] There are a number of clinical trials focused on the impact of physical activity and/or dietary modifications on ovarian cancer (LIVES - The Lifestyle Intervention for Ovarian Cancer Enhanced Survival), colon cancer (CHALLENGE - The Colon Health and Life-Long Exercise Change), prostate cancer (INTERVAL-GAP4 - Intense Exercise for Survival among Men with Metastatic Castrate-Resistant Prostate Cancer), and breast cancer (BWEL - The Breast Cancer Weight Loss).[12-15] A meta-analysis estimated that each 15 metabolic equivalent task-hour per week increase in physical activity after colorectal cancer diagnosis was associated with a 38% lower risk of mortality.[9]

The science behind beneficial effect of exercise in cancer subjects: There are multiple mechanisms cited for how exercise produces its beneficial effects, including through hormones, dopamine, transforming growth factor-B1 (TGF-B1), insulin-like growth factors (IGFs), microphthalmia/transcription factor E (MiT/TFE), mammalian target of rapamycin (mTOR), and secreted protein and rich in cysteine (SPARC). It has been shown in in-vitro and mice models that exercise inhibits cancer cell proliferation (for moderate- and high-intensity exercise, not low-intensity exercise) and induces apoptosis. One such mechanism involves dopamine release in the prefrontal cortex, serum, and cancer tissues. Dopamine binds to the dopamine receptor 2 (D2) upregulating the kinase phosphorylation and TGF-B1 to inhibit cancer cell proliferation.[10] Another mechanism involves IGFs which regulate mitosis and anti-apoptosis and affect proliferation and differentiation of cancer cells. Studies have shown that postmenopausal women have decreased IGF-1 and IGF-3 after walking training for 6 months, which inhibits IGF's anti-apoptosis effect in breast cancer, for example. Weight loss also reduces levels of IGF-1. Exercise induces skeletal muscle to produce SPARC, which promotes cleavage of caspase-3 and caspace-8, promoting cell apoptosis and inhibiting colon cancer. AMP activated protein kinase (AMPK) is an important center of homeostasis and regulator of mTOR kinase activity. In a mouse study involving hepatocarcinoma, exercise reduced the activity of mTOR kinase by stimulating AMPK, thereby reducing cancer cell proliferation. Finally, exercise can regulate cancer metabolism by inhibiting Warburg anaerobic glycolysis and weakening the hypoxia microenvironment of cancer. Lactic acid is the most important metabolite of glycolysis and cancer cells produce lots of lactic acid, creating a low-pH environment. Lactic acid suppresses the immune response, inhibiting T cells. Therefore, by inhibiting anaerobic glycolysis, exercise suppresses lactic acid production, improving the immune response to target cancer cells.[11] Additionally, exercise stimulates the activity of NK cell function, decreasing inflammation, enhancing antigen presentation, and mitigating the accumulation of aging cells in the elderly.[12]

Guidelines regarding exercise in cancer subjects and survivors: Both the American Cancer Society (ACS) and National Comprehensive Cancer Network (NCCN) have recommendations for cancer survivors regarding maintaining healthy weight and exercise among cancer survivors. [13,14].

The NCCN recommends:

* Be physically active every day - routine activities, recreation, or exercise
* Avoid being inactive for long periods each day
* Increase your heart rate each week: moderate-intensity activity for at least 150 to 300 minutes a week or vigorous-intensity activity for 75 minutes a week or a mix of moderate and vigorous-intensity activity
* Strengthen major muscles with resistance training 2 to 3 times a week
* Stretch major muscles on at least 2 of the days of high-intensity activity
* Healthy eating: focus on plant-based diet and limiting animal proteins such as red meat. Limiting processed foods.

The ACS recommends:

* Getting 150-300 minutes of moderate intensity or 75-150 minutes of vigorous intensity activity each week. Getting to or exceeding the upper limit of 300 minutes is ideal.
* Limit sedentary behavior such as sitting, lying down, watching TV, and other forms of screen-based entertainment.
* Healthy eating patterns
* Foods that are high in nutrients in amounts that help you get to and stay at a healthy body weight
* A variety of vegetables - dark green, red and orange, fiber-rich legumes and others
* Fruits, especially whole fruits in a variety of colors
* Whole grains
* Limiting red and processed meats, sugar-sweetened beverages, highly processed foods and refined grain products.

However, no clinical trials were found in our literature search that involve lung cancer subjects. There have been many articles describing the benefits of exercise for lung cancer survivors. Physical fitness, such as cardiorespiratory endurance and muscular strength have been independent predictors of survival.[15] However, the potential impact of exercise in lung cancer has not been fully explored and there are no guidelines for specific exercise programs. Avancini et al. proposed that a collaboration of exercise specialists is urgently needed to develop tailored programs based on subjects' needs, preferences and physical and psychological status.

It is becoming generally agreed that exercise improves oncological outcomes in cancer survivors. However, implementing programs for oncology rehabilitation have not been fully delineated. It has been proposed for oncology rehabilitation to piggy-back onto widely available exercise programs, such as cardiac rehabilitation.[16] It has also been proposed to use LIVESTRONG programs at the YMCA.[5] In a systematic review of sixteen randomized controlled trials including 2,684 participants, it was shown that the exercise programs that are most effective use technology-supported self-guided interventions.[17] Additionally, in a meta-analysis of 34 RCTs, exercise effects on quality of life and physical function were significantly improved with supervised rather than unsupervised exercise interventions.[18] Despite clear benefits, compliance with exercise program amongst cancer survivors has been an obstacle. In a systematic review of breast cancer subjects, only 6 of 17 trials demonstrated that significant intervention effects were maintained.[19] The study recommended greater transparency in reporting interventions to help maintain exercise programs. It will be important to determine when to start an exercise program, whether at diagnosis, during treatment or sometime after treatment, with the understanding that exercise can be considered another form of treatment and prevention. As the survivorship pool increases, it will be important to educate subjects that exercise is an essential component of treatment and secondary prevention.

Physical fitness, such as cardiorespiratory endurance and muscular strength have been independent predictors of survival.[20] However, no clinical trials were found in our literature search that specifically targeted lung cancer subjects on active treatment. As such, the potential impact of exercise in lung cancer subjects has not been fully explored and there are no guidelines for specific exercise programs. Furthermore, optimal timing, assessment for readiness, exercise specifics, and mode of administration of programs for oncology rehabilitation have not been fully delineated.

Lung cancer as focus: Subjects with lung cancer have a high symptom burden, due to their underlying disease and comorbidities. Surgical resection (segmentectomy, lobectomy or pneumonectomy), thoracic radiation and systemic cancer treatment can further add to deconditioning and low exercise capacity. It can be theorized that physical and pulmonary rehabilitation can potentially benefit these subjects and improve outcomes. A metanalysis which included 6 clinical trials and 221 participants showed that exercise training may improve or delay the decline in exercise capacity and disease specific global (Health Related Quality of Life) HRQoL for adults with advanced lung cancer.[21] However, there was no significant effects of exercise training on dyspnea, fatigue, feelings of anxiety and depression, or lung function. As the authors noted, there was significant heterogeneity between the trials, all of which had too small a sample size to derive any definitive conclusions.

Small randomized controlled studies have shown that pulmonary pre-habilitation and rehabilitation improve post-operative outcomes, post-operative pulmonary function and HRQoL.[22] Similarly, subjects who are undergoing chemotherapy were shown to benefit from an exercise program.[23] Despite multiple studies showing benefit, exercise program is not typically included in the treatment plan of lung cancer subjects. This is because this intervention has several challenges. Some of these issues are listed below.

1. Lostistic issues related to creating a multidisciplinary team of physiatrists, pulmonologist, oncologists, and other specialists for every subject
2. Creating a tailored regimen that is appropriate for each subject
3. Creating and maintaining enthusiasm amongst to participate in an exercise program
4. Time constraints of a busy oncology practice
5. Barriers related to number of visits to outsubject rehab facility, especially for subjects who live far from the rehab center.
6. Physical and emotional stress resulting from cancer diagnosis and treatment.
7. Comorbidities

Rationale for Northwell Health: Northwell Health is the largest health care system in the region, caring for over 300 lung cancer subjects every year. With a cohesive multidisciplinary team, accrual for this study will not be difficult. The virtual platform and the hands-on support from the PM&R and Salaso team will make it easier for subjects to participate regardless of their ability to travel frequently to the cancer center, and level of comfort with virtual platform.

Northwell is collaborating with Salaso for this project. Salaso is a digital health technology company that has online, mobile and telehealth solutions enabling providers to 'prescribe' evidence-based exercise programs for patients to complete virtually. The ExerciseRx project has two components:

* Platform Feasibility: Evaluating the feasibility of incorporating the Salaso platform into clinician workflow and understanding overall utilization of the platform by subjects (e.g., frequency of use, user satisfaction). Salaso will provide access to their ExerciseRx virtual exercise platform to Northwell providers and subjects and provide the necessary technical support to facilitate training and onboarding to the platform.
* Clinical Outcomes: In addition to feasibility of the platform the Northwell oncology team seeks to evaluate clinical impact for lung cancer subjects. For example, this will include evaluating pulmonary function and conducting the Six minute walk test (6MWT) and Sit to Stand Test (STS) at baseline and at the 12 month end of the study.

  * The additional clinical components of the study are Investigator Initiated and are funded by Northwell's Cancer Institute.

The Salaso digital technology is already integrated with Northwell's EMR. Platform satisfaction and FACT-L quality of life questionnaires will be directly administered to subjects via RedCap or on paper.

The following measures have been taken to protect HIPAA compliance

1. Despite Salaso's integration with Northwell EMR, Salaso will not have access to identifiable subject data. Although data will be collected via the ExerciseRx application, Salaso will only retain de-identified aggregate information and they will share the aggregate information directly with AstraZeneca. Questionnaires will be collected via RedCap. Biostatistician will be able to access RedCap data without PHI for statistical analysis.
2. Salaso will also passively collect data on the utilization of ExerciseRx, such as time spent in the platform and number of video views, to be shared with Northwell and Astrazeneca quarterly.

Disclosure:

Northwell Holdings, the investment arm of Northwell Health has invested in Salaso. Salaso's platform is already being used through Northwell's employee benefits portal (myHealthBody) and by the neurology department at Northwell (ExerciseRx). Salaso's platform is currently integrated with Allscripts.

In addition, AstraZeneca, is funding the use of the Salaso platform with Northwell and lung cancer patients. AstraZeneca funding will be used by Salaso to support the following:

* Development of the evidence-based exercises for the lung cancer patient population
* Salaso on the ground resource to support the training and onboarding of providers and patients to the Salaso ExerciseRx platform
* Collecting de-identified data on patient use of the platform, e.g. how many patients downloaded the ExerciseRx app, how often the patients used the app etc. (there will be no sharing of patient identifiable data).

The following measures are being taken to mitigate any perceived or potential conflict of interest (COI) related to Northwell Holding's investment in Salaso:

1. This study is investigator initiated. None of the investigators have any financial interests in Salaso.
2. Salaso's exercise program will be provided with no direct cost to subjects or providers.
3. Disclosure of Northwell's holding in Salaso will be made in the subject consent forms as well as in the final publication of study results.
4. Updates regarding the study, whether positive of negative will be provided to IRB as per Northwell IRB policies.
5. All investigators will engage in good clinical practices (GCP) and follow Human Subjects Research Protection guidelines per their Collaborative Institutional Training Initiative (CITI) training.

ELIGIBILITY:
Inclusion Criteria:

(1) Adults aged 18 and older (2) Have an ECOG PS of 0-2 (3) Have the ability to provide informed consent (4) Have the ability to engage in a virtual exercise platform (5) Commit to all study procedures as per protocol (6) Are deemed appropriate for virtual exercise program by the PM&R team (7) English speaking (8) Subjects with non-small cell lung cancer who belong to any of the three cohorts: (i) Cohort A: Peri-operative (subjects starting neoadjuvant chemotherapy or within 4-8 weeks after curative-intent thoracic surgery which could be segmentectomy, lobectomy of pneumonectomy), irrespective of adjuvant treatment - expected recruitment: 15 subjects (ii) Cohort B: Subjects starting definitive chemotherapy and radiation for locally advanced cancer - expected recruitment: 15 subjects (iii) Cohort C: Subjects with stage IV metastatic non-small cell lung cancer irrespective of type of treatment- expected recruitment: 30 subjects

Exclusion Criteria:

1. Unable to render informed consent
2. No other current active malignancy (beside lung cancer) at time of enrollment
3. Any contraindication to participating physically in an exercise program
4. Pregnant or breastfeeding at the time of screening visit
5. Any of the following contraindications to exercise use: acute post-operative subjects (within 8 weeks of operation; subjects with extreme fatigue, anemia, or ataxia; and general cardiovascular and respiratory contraindications for an exercise regimen.
6. Lack of proficiency in English sufficient for comprehension of trial source documents including the protocol, consent, and questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Viability | 12 months
  Feasibility of enabling patients to utilize a virtual exercise program, as assessed by percentage of eligible subjects who agree to enroll in the program, and percentage of enrolees who complete the program. Our objective is to have 50% of those who enroll complete the program at 12-months.

SECONDARY OUTCOMES:
Patient Satistfaction | 12 months
  Level of satisfaction in the ExerciseRx program as assessed by the Patient Satisfaction questionnaires
Provider Satisfaction | 12 months
  Provider satisfaction as assessed by provider satisfaction questionnaire to oncologists and PM&R physicians to determine whether they will use this platform to manage subjects

OTHER OUTCOMES:
Functional improvement, objectively determined as 6MWT | 12 months
  Physical endurance as assessed by the Six minute walk test (6MWT, measured in meters)
Functional improvement, subjectively determined | 12 months
  Change or maintenance of HRQoL as determined by FACT-L questionnaire which is a 36 -item self-report instrument that measures multidimensional quality of life. Score range is 0-28 and the sum of the individual scores is multiplied by 7 and then divided by the number of items answered. The higher the score, the better the QOL.
Functional improvement, objectively determined as PFTs | 12 months
  Improvement or maintenance of pulmonary function (PFT) as measured by DLCO (cc of CO/sec/mm of Hg), FVC (measured in liters), FEV1 (measured in liters over 1 second)
Functional improvement, objectively determined as STS | 12 months
  Sit to Stand Test (STS) measured in seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Northwell Health, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All patient data will be stored securely in RedCap database. This is minimal risk where all protected health information (PHI) will be kept in a secure redcap database.
Supporting Information: Study Protocol
Time Frame: The data will become available June 2024 and will be available until June 2026.
Access Criteria: The data will be accessible by pre-selected members of the research and biostatistics team, as well as the technology staff through RedCap which requires a user name, password and security authorization.
URL: https://redcap.northwell.edu/

REFERENCES:
- [Background] Miller KD, Nogueira L, Mariotto AB, Rowland JH, Yabroff KR, Alfano CM, Jemal A, Kramer JL, Siegel RL. Cancer treatment and survivorship statistics, 2019. CA Cancer J Clin. 2019 Sep;69(5):363-385. doi: 10.3322/caac.21565. Epub 2019 Jun 11. PMID 31184787
- [Background] Wang Q, Zhou W. Roles and molecular mechanisms of physical exercise in cancer prevention and treatment. J Sport Health Sci. 2021 Mar;10(2):201-210. doi: 10.1016/j.jshs.2020.07.008. Epub 2020 Jul 30. PMID 32738520
- [Background] Magne N, Melis A, Chargari C, Castadot P, Guichard JB, Barani D, Nourissat A, Largillier R, Jacquin JP, Chauvin F, Merrouche Y. Recommendations for a lifestyle which could prevent breast cancer and its relapse: physical activity and dietetic aspects. Crit Rev Oncol Hematol. 2011 Dec;80(3):450-9. doi: 10.1016/j.critrevonc.2011.01.013. Epub 2011 Feb 21. PMID 21334920
- [Background] Dennett AM, Sarkies M, Shields N, Peiris CL, Williams C, Taylor NF. Multidisciplinary, exercise-based oncology rehabilitation programs improve patient outcomes but their effects on healthcare service-level outcomes remain uncertain: a systematic review. J Physiother. 2021 Jan;67(1):12-26. doi: 10.1016/j.jphys.2020.12.008. Epub 2020 Dec 24. PMID 33358544
- [Background] Meyerhardt JA, Heseltine D, Niedzwiecki D, Hollis D, Saltz LB, Mayer RJ, Thomas J, Nelson H, Whittom R, Hantel A, Schilsky RL, Fuchs CS. Impact of physical activity on cancer recurrence and survival in patients with stage III colon cancer: findings from CALGB 89803. J Clin Oncol. 2006 Aug 1;24(22):3535-41. doi: 10.1200/JCO.2006.06.0863. Epub 2006 Jul 5. PMID 16822843
- [Background] Brown JC, Ligibel JA. Putting Exercise Into Oncology Practice: State-of-the-Science, Innovation, and Future Directions. Cancer J. 2019 Sep/Oct;25(5):316-319. doi: 10.1097/PPO.0000000000000397. PMID 31567458
- [Background] van Dam RM, Li T, Spiegelman D, Franco OH, Hu FB. Combined impact of lifestyle factors on mortality: prospective cohort study in US women. BMJ. 2008 Sep 16;337:a1440. doi: 10.1136/bmj.a1440. PMID 18796495
- [Background] Friedenreich CM, Neilson HK, Farris MS, Courneya KS. Physical Activity and Cancer Outcomes: A Precision Medicine Approach. Clin Cancer Res. 2016 Oct 1;22(19):4766-4775. doi: 10.1158/1078-0432.CCR-16-0067. Epub 2016 Jul 12. PMID 27407093
- [Background] Van Blarigan EL, Meyerhardt JA. Role of physical activity and diet after colorectal cancer diagnosis. J Clin Oncol. 2015 Jun 1;33(16):1825-34. doi: 10.1200/JCO.2014.59.7799. Epub 2015 Apr 27. PMID 25918293
- [Background] Zhang QB, Zhang BH, Zhang KZ, Meng XT, Jia QA, Zhang QB, Bu Y, Zhu XD, Ma DN, Ye BG, Zhang N, Ren ZG, Sun HC, Tang ZY. Moderate swimming suppressed the growth and metastasis of the transplanted liver cancer in mice model: with reference to nervous system. Oncogene. 2016 Aug 4;35(31):4122-31. doi: 10.1038/onc.2015.484. Epub 2015 Dec 21. PMID 26686088
- [Background] Renner K, Singer K, Koehl GE, Geissler EK, Peter K, Siska PJ, Kreutz M. Metabolic Hallmarks of Tumor and Immune Cells in the Tumor Microenvironment. Front Immunol. 2017 Mar 8;8:248. doi: 10.3389/fimmu.2017.00248. eCollection 2017. PMID 28337200
- [Background] Bigley AB, Spielmann G, LaVoy EC, Simpson RJ. Can exercise-related improvements in immunity influence cancer prevention and prognosis in the elderly? Maturitas. 2013 Sep;76(1):51-6. doi: 10.1016/j.maturitas.2013.06.010. Epub 2013 Jul 17. PMID 23870832
- [Background] NCCN Guidelines for Subjects Survivorship Care for Healthy Living 2020. https://www.nccn.org/subjects/guidelines/content/PDF/survivorship-hl-subject.pdf
- [Background] https://www.cancer.org/healthy/eat-healthy-get-active/acs-guidelines-nutrition-physical-activity-cancer-prevention/guidelines.htm
- [Background] Avancini A, Sartori G, Gkountakos A, Casali M, Trestini I, Tregnago D, Bria E, Jones LW, Milella M, Lanza M, Pilotto S. Physical Activity and Exercise in Lung Cancer Care: Will Promises Be Fulfilled? Oncologist. 2020 Mar;25(3):e555-e569. doi: 10.1634/theoncologist.2019-0463. Epub 2019 Nov 26. PMID 32162811
- [Background] Dittus KL, Lakoski SG, Savage PD, Kokinda N, Toth M, Stevens D, Woods K, O'Brien P, Ades PA. Exercise-based oncology rehabilitation: leveraging the cardiac rehabilitation model. J Cardiopulm Rehabil Prev. 2015 Mar-Apr;35(2):130-9. doi: 10.1097/HCR.0000000000000091. PMID 25407596
- [Background] Kiss N, Baguley BJ, Ball K, Daly RM, Fraser SF, Granger CL, Ugalde A. Technology-Supported Self-Guided Nutrition and Physical Activity Interventions for Adults With Cancer: Systematic Review. JMIR Mhealth Uhealth. 2019 Feb 12;7(2):e12281. doi: 10.2196/12281. PMID 30747720
- [Background] Buffart LM, Kalter J, Sweegers MG, Courneya KS, Newton RU, Aaronson NK, Jacobsen PB, May AM, Galvao DA, Chinapaw MJ, Steindorf K, Irwin ML, Stuiver MM, Hayes S, Griffith KA, Lucia A, Mesters I, van Weert E, Knoop H, Goedendorp MM, Mutrie N, Daley AJ, McConnachie A, Bohus M, Thorsen L, Schulz KH, Short CE, James EL, Plotnikoff RC, Arbane G, Schmidt ME, Potthoff K, van Beurden M, Oldenburg HS, Sonke GS, van Harten WH, Garrod R, Schmitz KH, Winters-Stone KM, Velthuis MJ, Taaffe DR, van Mechelen W, Kersten MJ, Nollet F, Wenzel J, Wiskemann J, Verdonck-de Leeuw IM, Brug J. Effects and moderators of exercise on quality of life and physical function in patients with cancer: An individual patient data meta-analysis of 34 RCTs. Cancer Treat Rev. 2017 Jan;52:91-104. doi: 10.1016/j.ctrv.2016.11.010. Epub 2016 Dec 5. PMID 28006694
- [Background] Abdin S, Lavallee JF, Faulkner J, Husted M. A systematic review of the effectiveness of physical activity interventions in adults with breast cancer by physical activity type and mode of participation. Psychooncology. 2019 Jul;28(7):1381-1393. doi: 10.1002/pon.5101. Epub 2019 May 15. PMID 31041830
- [Background] Peddle-McIntyre CJ, Singh F, Thomas R, Newton RU, Galvao DA, Cavalheri V. Exercise training for advanced lung cancer. Cochrane Database Syst Rev. 2019 Feb 11;2(2):CD012685. doi: 10.1002/14651858.CD012685.pub2. PMID 30741408
- [Background] Spruit MA. Pulmonary rehabilitation. Eur Respir Rev. 2014 Mar 1;23(131):55-63. doi: 10.1183/09059180.00008013. PMID 24591662
- [Background] Mustian KM, Sprod LK, Janelsins M, Peppone LJ, Mohile S. Exercise Recommendations for Cancer-Related Fatigue, Cognitive Impairment, Sleep problems, Depression, Pain, Anxiety, and Physical Dysfunction: A Review. Oncol Hematol Rev. 2012;8(2):81-88. doi: 10.17925/ohr.2012.08.2.81. PMID 23667857